CLINICAL TRIAL: NCT00438594
Title: Age 9 Follow-up of Preventive Intervention
Brief Title: Age 9 Follow-up of Preventive Intervention (Denver)
Acronym: DenverY09
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: U.S. Department of Justice (U.S. Federal Agency); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 03-0776; R01MH069891 (NIH)
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Child Rearing; Risk Reduction Behavior; Reproductive Behavior
Keywords: nurse; paraprofessional; home visits; pregnancy; welfare; child development
MeSH Terms: conditions — Risk Reduction Behavior; Reproductive Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (No Intervention): Control group
- Paraprofessional home visits (Experimental): home visitation by Paraprofessional
  Interventions: Behavioral: home visitation
- Nurse home visits (Experimental): home visitation by Nurse
  Interventions: Behavioral: home visitation

INTERVENTIONS:
Behavioral: home visitation — Home visits from mid-pregnancy until child age 2. Group 2 is visits by a paraprofessional; group 3 is visits by nurses.
  Arms: Nurse home visits; Paraprofessional home visits

SUMMARY:
To examine the impact of prenatal and infancy home visiting by paraprofessionals and by nurses from child age 2 through 9.

DETAILED DESCRIPTION:
This project supports a 9-year follow-up of 650 children and their families who were enrolled in a randomized trial of prenatal and infancy home visiting by paraprofessionals and by nurses; participating families were assigned to control, paraprofessional-, or nurse-visited conditions. Earlier phases of assessment found significant benefits for nurse- and paraprofessional-visited families and children, although the nurse effects tended to be larger. The current phase of follow-up is designed to determine whether the effects of the nurse and paraprofessional programs endure and grow through the child age 9.5.

The project is organized around seven questions:

1. Do the programs of nurse and paraprofessional home-visiting produce enduring effects on: a) mothers' life-course; b) qualities of care parents provide to their children; c) children's early-onset behavior problems; d) children's incoherence and aggression/destruction in response to story stems; e) children's executive, language, and intellectual functioning and school achievement?
2. To what extent are the beneficial effects of the programs on parental care-giving and children's development concentrated on those born to mothers with few psychological resources?
3. To what extent are the benefits of the programs on mothers and children equivalent for Mexican- Americans and European-Americans?
4. To what extent are the effects of the programs on antisocial behavior concentrated on boys? 5. To what extent are program effects moderated by school and neighborhood contexts?

6. To what extent are the effects of the programs on children's development explained by impacts of the programs on women's prenatal smoking, maternal life-course, qualities of parental caregiving, and children's earlier language development, executive functioning, and emotional regulation? 7. To what extent are the initial costs of the programs recovered in reduced expenditures for other government services during the first nine years of the first child's life?

ELIGIBILITY:
Inclusion Criteria:

* Women from 21 antepartum clinics serving low-income women in Denver recruited if they had no previous live births and either qualified for Medicaid or had no private insurance.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2004-02; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
fewer subsequent pregnancies | When first child is 9
increased interval between the birth of the first and second child | When first child is 9
reduced use of welfare | When first child is 9
increased participation in the work force | When first child is 9
reduced behavioral problems due to use of alcohol and drugs | When first child is 9
fewer arrests | When first child is 9
increased qualities of care parents provide to their children as reflected in fewer verified reports of child abuse and neglect and observations of coercive mother-child interaction. | When first child is 9
children's early-onset behavior problems (both externalizing and internalizing) reported by parents and teachers at home, at school, and with peers. | At child age 9
children's aggressive and destructive themes and narrative coherence in their responses to story stems. | At child age 9
executive functions and school achievement. | At child age 9

CONTACTS AND LOCATIONS:
Overall Officials: David L Olds, PhD, Principal Investigator — University of Colorado, Denver

REFERENCES:
- [Background] Olds DL, Robinson J, O'Brien R, Luckey DW, Pettitt LM, Henderson CR Jr, Ng RK, Sheff KL, Korfmacher J, Hiatt S, Talmi A. Home visiting by paraprofessionals and by nurses: a randomized, controlled trial. Pediatrics. 2002 Sep;110(3):486-96. doi: 10.1542/peds.110.3.486. PMID 12205249
- [Background] Olds DL, Robinson J, Pettitt L, Luckey DW, Holmberg J, Ng RK, Isacks K, Sheff K, Henderson CR Jr. Effects of home visits by paraprofessionals and by nurses: age 4 follow-up results of a randomized trial. Pediatrics. 2004 Dec;114(6):1560-8. doi: 10.1542/peds.2004-0961. PMID 15574615
- [Derived] Olds DL, Holmberg JR, Donelan-McCall N, Luckey DW, Knudtson MD, Robinson J. Effects of home visits by paraprofessionals and by nurses on children: follow-up of a randomized trial at ages 6 and 9 years. JAMA Pediatr. 2014 Feb;168(2):114-21. doi: 10.1001/jamapediatrics.2013.3817. PMID 24296904